CLINICAL TRIAL: NCT06172114
Title: Bovine-derived Xenograft (Bio-Oss Collagen) With or Without Leukocyte-platelet Rich Fibrin (L-PRF) for Alveolar Ridge Preservation After Tooth Extraction: a Randomized Controlled Trial
Brief Title: Bovine-derived Xenograft With or Without L-PRF for Alveolar Ridge Preservation After Tooth Extraction: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Abeer Hakam, Assistant professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MBRU-PRF
Record Dates: First submitted 2023-11-22; First posted 2023-12-15 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Dental Implants; Tooth Extraction; Bone Regeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (C) (Active Comparator): Xenograft + resorbable collagen membrane
  Interventions: Procedure: Alveolar ridge preservation using sticky bone
- Test group (T) (Experimental): Xenograft combined with L-PRF + resorbable collagen membrane
  Interventions: Procedure: Alveolar ridge preservation using sticky bone

INTERVENTIONS:
Procedure: Alveolar ridge preservation using sticky bone — In the test group the xenograft will be mixed in with the L-PRF then placed into the socket.

SUMMARY:
The study is prospective randomized clinical trial that aims to evaluate the adjunctive use of L-PRF in promoting the desired vascularization and bone fill in small and large defects following tooth extraction and report on the long-term implant and patient outcomes

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over.
* Require extraction of anterior or posterior single tooth due to caries, endodontic and prosthetic complications.
* The tooth that requires extraction is bordered by two teeth.
* Controlled oral hygiene (full-mouth plaque and bleeding scores ≤ 25% at baseline).
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent.

Exclusion Criteria:

* Localised / generalised periodontitis.
* Presence of acute periapical lesion.
* Bone metabolic disease and/or taking medications that affect bone metabolism.
* Long term use of non-steroidal anti-inflammatory medications.
* History of malignancy, radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Severe bruxism or parafunctional habits.
* Large occlusal discrepancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Implant survival / success rate will be assessed clinically after one year of implant restoration and annually up to three years. | 2 years
Patient postoperative experience will be assessed using visual analogue scale during the first week following tooth extraction and ridge preservation. | 2 years
  Reporting a score will be done using the pain visual analogue scale. Minimum value is 0 which is no pain and maximum value is 10 which is the worst pain ever experienced.

SECONDARY OUTCOMES:
Changes in width and height of alveolar ridge will be assessed at the time of tooth extraction and ridge preservation, six months (prior to implant placement) and annually up to two years using cone beam computed tomography (CBCT). | 2 years
Need for additional bone augmentation will only be assessed at the time of implant placement by recording the use of bone graft (if required) in the clinical notes. | 2 years
Changes in peri-implant marginal bone level will be assessed at implant placement (baseline) and after one year of implant restoration and annually up to two years using standardized peri-apical radiograph. | 2 years
Soft tissue levels (midbuccal marginal tissue level changes, interproximal papilla level changes and changes in width of keratinised tissue) will be assessed at implant placement (baseline), at 1 year and at 2 years | 2 years
Biological complications (i.e. peri-implant diseases) will be assessed clinically using periodontal probe after one year of implant restoration and annually up to two years. | 2 years

IPD SHARING:
Plan to Share IPD: No